CLINICAL TRIAL: NCT04405128
Title: Brain TV (Tissue Velocimetry) for Emergency Assessment of Suspected Stroke
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: Nihon Kohden (Industry)
Responsible Party: Sponsor
Other Study IDs: 0679
Record Dates: First submitted 2020-05-20; First posted 2020-05-28 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2021-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transcranial Tissue Doppler (TCTD) — Doppler ultrasound technique called "Brain Tissue Velocimetry" (Brain TV), to investigate brain tissue motion over the cardiac cycle.
Diagnostic Test: Brain Magnetic Resonance Imaging — Brain MRI for investigation of brain tissue motion in the presence of suspected stroke.

SUMMARY:
This study uses a Doppler ultrasound technique being developed at the University of Leicester called "Brain Tissue Velocimetry" (Brain TV), to investigate brain tissue motion over the cardiac cycle.

DETAILED DESCRIPTION:
Brain motion is highly sensitive to heart and brain biomechanics, but the impact of brain injury on brain tissue motion has yet to be explored. Preliminary brain tissue motion measurements from a small number of patients suggest that brain biomechanics may be disturbed in the presence of brain injury. This study combines transcranial tissue Doppler (TCTD) ultrasound with brain magnetic resonance imaging (MRI) to establish whether analysis of brain tissue motion provides clinically useful information for emergency diagnosis and monitoring of suspected stroke.

ELIGIBILITY:
Inclusion Criteria:

* Participant (or consultee) is willing and able to give informed consent (or assent) for participation in the study.
* Adult, aged 18 years or over.
* Suspected stroke (any severity and any stroke type).

Exclusion Criteria:

* Unable (in the investigators' opinion), or unwilling, to comply with the study requirements.
* Patients with pre-existing chronic brain conditions that may make affect informed consent, such as severe learning difficulties, dementia, or Alzheimer's disease, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with suspected stroke will be identified and recruited by the Emergency Department (ED) research team and/or members of the direct care team within the Hyper Acute Stroke Unit (HASU).
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
MRI measurement | Up to 5 days.
  This study will perform brain MRI for brain tissue motion for selective patients with suspected stroke.
TCTD measurement | Up to 5 days.
  The study will generate a library of Brain TV measurements for exploratory (descriptive) analysis and imaging of brain tissue pulsations in patients with suspected stroke to evaluate the potential for clinical device development.

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Chung, PhD, Principal Investigator — King's College, London
Locations (1):
- University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided